CLINICAL TRIAL: NCT02941705
Title: Regress-HFpEF: Regression of Fibrosis & Reversal of Diastolic Dysfunction in HFpEF Patients Treated With Allogeneic CDCs
Brief Title: Regression of Fibrosis & Reversal of Diastolic Dysfunction in HFpEF Patients Treated With Allogeneic CDCs
Acronym: RegressHFpEF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Eduardo Marbán, MD, PhD, Director, Heart Institute, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 54823
Record Dates: First submitted 2016-08-10; First posted 2016-10-21 (Estimated); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Congestive Heart Failure; Heart Failure, Diastolic
Keywords: stem cell research
MeSH Terms: conditions — Heart Failure; Heart Failure, Diastolic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RECIEVED CELLS (Active Comparator): this arm will receive the CDCs /CAP 1002 solution
  Interventions: Biological: Allogeneic Derived Cells
- CONTROL ARM (Placebo Comparator): this arm will receive a solution during randomization but will not receive the CDCs
  Interventions: Biological: Placebo/Control Arm

INTERVENTIONS:
Biological: Allogeneic Derived Cells — patients will have the CAP-1002 solution delivered through a coronary catheter inserted in the right and left coronary arteries using standard techniques in the cardiac catheterization laboratory. A right heart catheter will be used to obtain baseline (pre-infusion) hemodynamics.
  Other Names: CAP-1002
  Arms: RECIEVED CELLS
Biological: Placebo/Control Arm — patients will receive the placebo through a coronary catheter inserted in the right and left coronary arteries using standard techniques in the cardiac catheterization laboratory. A right heart catheter will be used to obtain baseline (pre-infusion) hemodynamics.
  Other Names: Placebo
  Arms: CONTROL ARM

SUMMARY:
Perform a randomized, double blind, placebo-controlled Phase 2a feasibility study to determine whether treatment of HFpEF patients with intracoronary allogeneic CDCs affects clinical functional status (QOL scores), exercise tolerance (6MHW), exercise hemodynamics (supine exercise ergometry during right heart catheterization), myocardial interstitial fibrosis (MRI with native T1 mapping and calculation of extracellular volume [ECV] after gadolinium administration), macroscopic fibrosis by delayed gadolinium enhancement (DGE), and diastolic function (catheterization, echocardiography, BNP).

Treatment of patients with symptomatic hypertensive heart disease-induced HFpEF with allogeneic CDCs will be safe and will improve clinical functional status, exercise tolerance/hemodynamics, myocardial interstitial structure, and diastolic function; the mechanisms underlying these improvements will be reflected in changes in plasma biomarkers that indicate a reduction in pro-inflammatory and pro-fibrotic signaling.

DETAILED DESCRIPTION:
Heart failure with Preserved Ejection Fraction (HFpEF) is a distinct clinical heart failure syndrome and represents a critical unmet need in cardiovascular medicine. HFpEF patients have a marked increase in morbidity and mortality and a profound clinical disability. However, to date, no management strategies have been demonstrated to decrease morbidity and mortality or decrease the clinical disability suffered by HFpEF patients. Investigators have postulated that one pivotal reason that previous randomized clinical studies have failed to show efficacy in HFpEF trials centers around the incomplete understanding of the pathophysiologic mechanisms underlying the development of HFpEF. Studies in Veteran patients with HFpEFand in relevant animal models of HFpEF have demonstrated that one critical mechanism contributing to HFpEF are changes in the cardiac interstitium and extracellular matrix (ECM) fibrillar collagen homeostasis. Preliminary studies presented in this application demonstrate that a highly novel application of stem cell therapy to a rodent model of HFpEF results in regression of ECM fibrosis and reversal of LV diastolic dysfunction. These preliminary studies form the foundation for the 3 specific aims proposed in this application that targets HFpEF in Veterans.

The primary and secondary objectives of this study are too determine the safety profile of CAP-1002 administered by intracoronary infusion in patients with Heart Failure and a Preserved Ejection Fraction (HFpEF) and to assess exploratory efficacy endpoints to determine whether treatment of HFpEF patients with intracoronary allogeneic CDCs affects clinical functional status (QOL scores), exercise tolerance (6 Minute Walk Test - 6MWT), exercise hemodynamics (supine exercise ergometry during right heart catheterization), myocardial interstitial fibrosis (MRI with native T1 mapping and calculation of extracellular volume [ECV] after gadolinium administration), macroscopic fibrosis by delayed gadolinium enhancement (DGE), and diastolic function (catheterization, echocardiography, BNP).

If a patient fulfills the inclusion criteria of clinical HF, preserved EF, increased BNP, and increased LA size and has none of the exclusion criteria (see details below), they will be consented and undergo CT coronary angiography (to define the coronary anatomy) and donor-specific antibodies (DSA) screen. If significant CAD is identified by CT and confirmed by subsequent coronary arteriography and FFR, subjects will be referred to their physician for consideration of a revascularization procedure. If such subjects undergo a revascularization procedure, subjects may be reconsidered and rescreened for the study, minus a repeat CT, after a minimum of 3 months post-revascularization.

All patients will have CAP-1002 or placebo delivered through a coronary catheter inserted in the right and left coronary arteries using standard techniques in the cardiac catheterization laboratory. A right heart catheter will be used to obtain baseline (pre-infusion) hemodynamics. All patients will receive 25 million cells (CAP-1002) or placebo in each of the 3 coronary arteries. Sequential dose administration of 25 million cells each suspended in10 mL of cryopreservation solution (CryoStor® CS10, BioLife Solutions, Inc.) containing 10% dimethyl sulfoxide (DMSO), and 1800 units heparin and 45 mcg nitro will be delivered via a coronary artery catheter. Additionally, four milliliters of an intermediate wash solution containing saline is also administered to each patient. Patients randomized to the placebo group will receive placebo injections consisting of CAP-1002 minus the active CDC constituent. Each 10ml bag of 25 million cells will be infused over 1 ml/min. All procedures will be performed by the cardiac interventionist (Dr Fernandes). The patient will receive local anesthesia +/- gentle conscious sedation if undue anxiety. During and in between infusions, multiple measures of gas exchange, hemodynamics, including blood pressure and heart rate and monitoring for any arrhythmias (ventricular and supra-ventricular). Fluids are permitted for hypotension during the procedure, as are low dose inotropes such as dobutamine and use of inhaled nitric oxide. VPCs or NSVT can be seen with insertion of the PA catheter as it traverses the RV and is easily remedied by catheter withdrawal. Oxygen will be used in those patients already on O2 therapy at baseline and if needed to treat temporary hypoxia should this occur. If significant adverse events occur, the cell infusion will be terminated. Pre-specified infusion related events include the following within 6 hours of CDC infusion: refractory hypotension requiring pressors and inotropes, significant hypoxemia requiring FiO2 > 0.4 or an increment of > 0.2 from baseline, new cardiac arrhythmia requiring cardioversion, ventricular tachycardia, ventricular fibrillation, asystole or pulseless electrical activity, acute severe transfusion reaction (immune or infection related).

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 50 years old, male or female
2. LVEF ≥ 50%
3. Symptoms and physical findings of chronic heart failure (NYHA class II- ambulatory IV)
4. Treatment with a stable, maximally-tolerated dose of diuretic(s) for a minimum of 30 days prior to randomization.
5. Left atrial (LA) enlargement defined by at least one of the following: LA width (diameter) ≥ 3.8 cm or LA length ≥ 5.0 cm or LA area ≥ 20 cm2 or LA volume ≥ 55 mL or LA volume index ≥ 29 mL/m2
6. BNP > 125 pg/ml for patients in NSR or > 150 pg/ml for patients in AF (BNP are BMI corrected) or resting PCWP > 15 mmHg, or exercise PCWP > 18 mmHg

Exclusion criteria-Specific to HFpEF

1. Any prior echocardiographic measurement of LVEF < 40 %
2. Acute coronary syndrome (including MI), cardiac surgery, other major CV surgery, or percutaneous coronary intervention (PCI) within the 3 months prior to randomization
3. Unrevascularized, hemodynamically significant CAD (FFR < 0.75)
4. Current acute decompensated HF
5. Alternative diagnoses that in the opinion of the investigator could account for the patient's HF symptoms (i.e., dyspnea, fatigue) such as severe pulmonary disease (i.e., requiring home oxygen, chronic nebulizer therapy, chronic oral steroid therapy); hemoglobin (Hgb) < 10 g/dl; body mass index (BMI) > 40 kg/m2
6. Use of investigational drugs or treatments at the time of enrollment
7. Systolic blood pressure > 150 mmHg but < 180 mmHg unless receiving 3 or more antihypertensive drugs
8. History of any dilated cardiomyopathy; right sided HF in the absence of left-sided structural heart disease; Pericardial constriction, genetic hypertrophic cardiomyopathy, or infiltrative cardiomyopathy; clinically significant congenital heart disease; hemodynamically significant valvular heart disease
9. Stroke, transient ischemic attack, carotid surgery or carotid angioplasty within the 3 months
10. Uncontrolled dysrhythmia; symptomatic or sustained ventricular tachycardia or atrial fibrillation or flutter with a resting ventricular rate > 110 beats per minute (bpm)
11. Prior major organ transplant or intent to transplant (i.e., on transplant list)
12. Hepatic disease as determined by any one of the following: SGOT (AST) or SGPT (ALT) values exceeding 3x the upper limit of normal (ULN), bilirubin > 1.5 mg/dl; history of chronic viral hepatitis
13. Chronic Kidney Disease with eGFR < 30 mL/min/1.73 m2; serum potassium > 5.5 mmol/L (mEq/L)
14. History or presence of any other disease with a life expectancy of < 3 years
15. Non-compliance to medical regimens
16. Drug or alcohol abuse within the last 12 months
17. History of malignancy within the past 5 years
18. Pregnant or nursing (lactating) women confirmed by a positive human chorionic gonadotropin (hCG); women of child-bearing potential (physiologically capable of becoming pregnant), unless using highly effective contraception methods during study

Exclusion criteria-Specific to CAP-1002 (not listed above)

1. Diagnosis of active myocarditis
2. Known hypersensitivity to contrast agents or previous H/O HIT
3. Known hypersensitivity to dimethyl sulfoxide (DMSO)
4. Known hypersensitivity to bovine products
5. Active infection not responsive to treatment
6. Active allergic reactions, connective tissue diseases or autoimmune disorders
7. History of cardiac tumor or cardiac tumor demonstrated on screening
8. History of previous stem cell therapy
9. History of treatment with immunosuppressive agents, including chronic systemic corticosteroids, biologic agents targeting the immune system, anti-tumor and anti-neoplastic drugs or anti-VEGF within 6 months prior to enrollment (not including drug-eluting coronary stents)
10. Human Immunodeficiency Virus (HIV) infection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zile, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The proposed goal in the DOD application was a sample size of 40 patients. The actual enrolled number was 27. We were unable to reach the goal of 40 due to constraints in time, budget, and patient availability. In part these constraints were exaggerated by the COVID 19 pandemic (declared 3-1-2020) which severely constrained enrollment in all clinical trials in the USA.
  2 subjects who were screen failures who were never consented. One was screened/enrolled but withdrew prior to cell infusion.
Period: Overall Study
Arm/Group | RECIEVED CELLS | CONTROL ARM
Started (We are defining 'started' as having been randomized to a treatment group. The three subjects who were screened but did not complete the study all withdrew prior to randomization. Two subjects were screen failures and one subject withdrew prior to randomization. Therefore, we have not included those individuals in the total number of subjects 'started' since they were never randomized to a treatment group.) | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RECIEVED CELLS | CONTROL ARM | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 8 | 8 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: the Safety Profile of CAP 1002; Any Subjects Experiencing Any Safety Related Events During or Post Intracoronary Delivery and During the Follow up Period.
Description: any subjects experiencing any safety related events during or post intracoronary delivery and during the follow up period.
  Safety outcomes will be measured through TIMI flow 0-2, acute myocarditis within one month of intracoronary infusion, ventricular tachycardia or ventricular fibrillation within 72 hours of intracoronary infusion, sudden unexpected death within 72 hours of intracoronary infusion defined as occurring 1 hour within in symptom onset or witnessed death in a subject previously observed to be well within the preceding 24 hours without an identified cause, or a major adverse cardiac event within 72 hours of intracoronary infusion.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | RECIEVED CELLS | CONTROL ARM
Number analyzed (Participants) | 13 | 13
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 1 year following infusion.
Arm/Group | RECIEVED CELLS | CONTROL ARM
All-Cause Mortality (participants affected / at risk) | 1/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13 | 3/13
Other Adverse Events (participants affected / at risk) | 12/13 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RECIEVED CELLS (N=13) | CONTROL ARM (N=13)
Ischemic Stroke (Vascular disorders) | 1 | 0
Vertigo/sinus infection (Ear and labyrinth disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 0
Chronotropic incompetence/ pacemaker implanted (Cardiac disorders) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Acute HFpEF exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pancreatic adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RECIEVED CELLS (N=13) | CONTROL ARM (N=13)
Acute Cystitis (Infections and infestations) | 0 (0) | 1 (1) — Acute Cystitis with Hematuria and Dyspnea
Acute HFpEF Exac (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
AKI (Renal and urinary disorders) | 1 (1) | 2 (2)
Anxiety during RHC (Nervous system disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 2 (2) | 1 (1)
Atrial Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Back Pain with Spinal Nerve Ablation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 4 (4) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (3) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Anemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — EGD for Anemia without Evidence of Bleed
Elevated Bilirubin (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Elevated BNP (Cardiac disorders) | 0 (0) | 1 (1)
Elevated Troponin (Cardiac disorders) | 7 (7) | 9 (9)
Emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — Ferumoxytol Infusion
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hypervolemia (Cardiac disorders) | 0 (0) | 3 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1)
Increased Swelling (Cardiac disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Ischemic Stroke (Vascular disorders) | 0 (0) | 1 (1)
Hypervolemia (Cardiac disorders) | 1 (1) | 0 (0) — IV Lasix for Volume Overload
Laryngeal papillomas excision (Gastrointestinal disorders) | 0 (0) | 1 (1)
Memory Loss (Nervous system disorders) | 1 (1) | 0 (0)
Nonflow Limiting Staining in Prox LCx (Cardiac disorders) | 1 (1) | 0 (0)
Pancreatic Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Potential Metabolic Acidosis (Endocrine disorders) | 0 (0) | 1 (1)
Right Knee Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin tear from blood pressure cuff (Surgical and medical procedures) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Syncopal Episode (Nervous system disorders) | 2 (2) | 0 (0)
Tachy Arrythmia (Cardiac disorders) | 0 (0) | 1 (1)
Thrombophebitis of Right Arm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Transaminitis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Transient AV Block during RCA infusion (Cardiac disorders) | 0 (0) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
UTI (Renal and urinary disorders) | 1 (1) | 0 (0)
Vertigo/Chronic Sinus Infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT02941705/Prot_SAP_001.pdf